CLINICAL TRIAL: NCT01275079
Title: Change of Nasalance After Tonsillectomy in Thai Adult
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Permpoon Piyaman, Department of Otolaryngology , Faculty of Medicine , Chulalongkorn University
Other Study IDs: Resident_Permpoon
Record Dates: First submitted 2010-11-26; First posted 2011-01-12 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Voice Quality; Tonsillectomy
Keywords: tonsillectomy; nasalance; tonsil volume; Thai; adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Rt. and Lt.tonsil
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to analyze the change of nasalance after tonsillectomy in Thai adults.

ELIGIBILITY:
Inclusion Criteria:

* Thai adults age over 18 years who were perform bilateral tonsillectomy
* The pathological are not malignancy

Exclusion Criteria:

* Craniofacial anomalies
* Neurological problems
* History of Peritonsillar abscess
* Performed other operation beside tonsillectomy
* Can't read Thais
* Visual problem that effect reading
* Nasal disease that cause nasal obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thai adults who were performed tonsillectomy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Permpoon Piyaman, MD, Principal Investigator — Department of otolaryngology, faculty of medicine, Chulalongkorn university
Locations (1):
- Department of otolaryngology, faculty of medicine, Chulalongkorn university, Bangkok, Bangkok, Thailand